CLINICAL TRIAL: NCT01254045
Title: Double-blind Placebo Controlled Study of Oxytocin in Fragile X Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Allan Reiss, Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SU-11182010-7215; 8618 (Other: Stanford University IRB eProtocol)
Record Dates: First submitted 2010-12-02; First posted 2010-12-06 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- placebo, oxytocin 24IU, oxytocin 48IU (Experimental): intranasal placebo (48 international units; 4IU per puff) once at baseline, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal oxytocin (24 international units; 4IU per puff) and intranasal placebo (24 international units; 4IU per puff) once at time 2, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal oxytocin (48 international units; 4IU per puff) once at time 3, 6 puffs (3 puffs per nostril) from each of 2 bottles
  Interventions: Drug: placebo; Drug: oxytocin 24IU; Drug: oxytocin 48IU
- oxytocin 24IU, placebo, oxytocin 48IU (Experimental): intranasal oxytocin (24 international units; 4IU per puff) and intranasal placebo (24 international units; 4IU per puff) once at baseline, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal placebo (48 international units; 4IU per puff) once at time 2, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal oxytocin (48 international units; 4IU per puff) once at time 3, 6 puffs (3 puffs per nostril) from each of 2 bottles
  Interventions: Drug: placebo; Drug: oxytocin 24IU; Drug: oxytocin 48IU
- oxytocin 48IU, oxytocin 24IU, placebo (Experimental): intranasal oxytocin (48 international units; 4IU per puff) once at baseline, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal oxytocin (24 international units; 4IU per puff) and intranasal placebo (24 international units; 4IU per puff) once at time 2, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal placebo (48 international units; 4IU per puff) once at time 3, 6 puffs (3 puffs per nostril) from each of 2 bottles
  Interventions: Drug: placebo; Drug: oxytocin 24IU; Drug: oxytocin 48IU
- oxytocin 24IU, oxytocin 48IU, placebo (Experimental): intranasal oxytocin (24 international units; 4IU per puff) and intranasal placebo (24 international units; 4IU per puff) once at baseline, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal oxytocin (48 international units; 4IU per puff) once at time 2, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal placebo (48 international units; 4IU per puff) once at time 3, 6 puffs (3 puffs per nostril) from each of 2 bottles
  Interventions: Drug: placebo; Drug: oxytocin 24IU; Drug: oxytocin 48IU
- oxytocin 48IU, placebo, oxytocin 24IU (Experimental): intranasal oxytocin (48 international units; 4IU per puff) once at baseline, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal placebo (48 international units; 4IU per puff) once at time 2, 6 puffs (3 puffs per nostril) from each of 2 bottles ; intranasal oxytocin (24 international units) and intranasal placebo (24 international units; 4IU per puff) once at time 3, 6 puffs (3 puffs per nostril) from each of 2 bottles
  Interventions: Drug: placebo; Drug: oxytocin 24IU; Drug: oxytocin 48IU
- placebo, oxytocin 48IU, oxytocin 24IU (Experimental): intranasal placebo (48 international units; 4IU per puff) once at baseline, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal oxytocin (48 international units; 4IU per puff) once at time 2, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal oxytocin (24 international units; 4IU per puff) and intranasal placebo (24 international units; 4IU per puff) once at time 3, 6 puffs (3 puffs per nostril) from each of 2 bottles
  Interventions: Drug: placebo; Drug: oxytocin 24IU; Drug: oxytocin 48IU

INTERVENTIONS:
Drug: placebo — intranasal placebo (48 international units)
Drug: oxytocin 24IU — intranasal oxytocin (24 international units) and intranasal placebo (24 international units)
  Other Names: Syntocinon
Drug: oxytocin 48IU — intranasal oxytocin (48 international units)
  Other Names: Syntocinon

SUMMARY:
The purpose of this study is to determine whether the medication oxytocin is an effective and tolerable treatment in adolescent males with fragile X syndrome (FraX) for improving socially appropriate behaviors and reducing social anxiety.

DETAILED DESCRIPTION:
Twelve male adolescent (13-24 years) subjects with confirmed genetic diagnosis of FraX (full mutation) will participate in this randomized double-blind placebo-controlled study. They will receive a dose of either 24 IU oxytocin, 48 IU oxytocin or placebo at each of three visits to the lab, with each visit spaced one week apart. The efficacy of each dose will be evaluated using behavioral, cognitive and physiological metrics. If individual subject results suggest that either of the oxytocin dosage levels (24 IU or 48 IU) is superior to placebo in the double-blind phase, a single-blind trial using the optimal dosage of oxytocin will then be administered daily for 14 days by parents at home. Subjects will then come into the lab for a final assessment on Day 30. Determination of beneficial response to oxytocin will be based on a 20% change (improvement) in behavior or test performance (see below). If both oxytocin dosage levels provide similar benefits compared to placebo, the lower dose will be chosen for the 14 day single-blind trial.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed genetic diagnosis of Fragile X (FraX) (full mutation).
2. Male (who have more serious effects due to the X chromosome nature of the disorder)
3. Age 13-29 years.
4. Parent of adolescent must be willing to sign informed consent.
5. Intelligence Quotient (IQ) > 42.

Exclusion Criteria:

1. Cardiac risk factors.
2. Medication exclusions: opiates or opiate antagonists, corticosteroids, typical or atypical antipsychotics.

Ages: 13 Years to 29 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2007-02; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan L Reiss, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Hall SS, Lightbody AA, McCarthy BE, Parker KJ, Reiss AL. Effects of intranasal oxytocin on social anxiety in males with fragile X syndrome. Psychoneuroendocrinology. 2012 Apr;37(4):509-18. doi: 10.1016/j.psyneuen.2011.07.020. Epub 2011 Aug 20. PMID 21862226

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Ten enrolled. One on antipsychotic mediation at baseline excluded, and one lost to follow-up after baseline. Eight participants included in data analysis. Each participant received a dose of either oxytocin(OT) 24 international units (IU)/intranasal placebo 24IU, OT 48IU, or placebo 48IU at each of 3 weekly visits.
Groups:
- Placebo 48IU, Oxytocin 24IU/Placebo 24IU, Oxytocin 48IU: intranasal placebo (48 international units; 4IU per puff) once at baseline, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal oxytocin (24 international units; 4IU per puff) and placebo (24 international units; 4IU per puff) once at time 2, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal oxytocin (48 international units; 4IU per puff) once at time 3, 6 puffs (3 puffs per nostril) from each of 2 bottles
- Oxytocin 24IU/Placebo 24IU, Placebo 48IU, Oxytocin 48IU: intranasal oxytocin (24 international units; 4IU per puff) and intranasal placebo (24 international units; 4IU per puff) once at baseline, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal placebo (48 international units; 4IU per puff) once at time 2, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal oxytocin (48 international units; 4IU per puff) once at time 3, 6 puffs (3 puffs per nostril) from each of 2 bottles
- Oxytocin 48IU, Oxytocin 24IU/Placebo 24IU, Placebo 48IU: intranasal oxytocin (48 international units; 4IU per puff) once at baseline, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal oxytocin (24 international units; 4IU per puff) and intranasal placebo (24 international units; 4IU per puff) once at time 2, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal placebo (48 international units; 4IU per puff) once at time 3, 6 puffs (3 puffs per nostril) from each of 2 bottles
- Oxytocin 24IU/Placebo 24IU, Oxytocin 48IU, Placebo 48IU: intranasal oxytocin (24 international units; 4IU per puff) and intranasal placebo (24 international units; 4IU per puff) once at baseline, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal oxytocin (48 international units; 4IU per puff) once at time 2, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal placebo (48 international units; 4IU per puff) once at time 3, 6 puffs (3 puffs per nostril) from each of 2 bottles
- Oxytocin 48IU, Placebo 48IU, Oxytocin 24IU/Placebo 24IU: intranasal oxytocin (48 international units; 4IU per puff) once at baseline, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal placebo (48 international units; 4IU per puff) once at time 2, 6 puffs (3 puffs per nostril) from each of 2 bottles ; intranasal oxytocin (24 international units; 4IU per puff) and intranasal placebo (24 international units; 4IU per puff) once at time 3, 6 puffs (3 puffs per nostril) from each of 2 bottles
- Placebo 48IU, Oxytocin 48IU, Oxytocin 24IU/Placebo 24IU: intranasal placebo (48 international units; 4IU per puff) once at baseline, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal oxytocin (48 international units; 4IU per puff) once at time 2, 6 puffs (3 puffs per nostril) from each of 2 bottles; intranasal oxytocin (24 international units; 4IU per puff) and intranasal placebo (24 international units; 4IU per puff) once at time 3, 6 puffs (3 puffs per nostril) from each of 2 bottles
Period: First/Baseline (1 Day at Week 1 )
Arm/Group | Placebo 48IU, Oxytocin 24IU/Placebo 24IU, Oxytocin 48IU | Oxytocin 24IU/Placebo 24IU, Placebo 48IU, Oxytocin 48IU | Oxytocin 48IU, Oxytocin 24IU/Placebo 24IU, Placebo 48IU | Oxytocin 24IU/Placebo 24IU, Oxytocin 48IU, Placebo 48IU | Oxytocin 48IU, Placebo 48IU, Oxytocin 24IU/Placebo 24IU | Placebo 48IU, Oxytocin 48IU, Oxytocin 24IU/Placebo 24IU
Started | 2 (One completed all baseline measures including administration of placebo, but then lost to follow-up.) | 2 | 2 | 1 | 1 | 1
Completed | 1 | 2 | 2 | 1 | 1 | 1
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Period: Second/Time 2 (1 Day at Week 2)
Arm/Group | Placebo 48IU, Oxytocin 24IU/Placebo 24IU, Oxytocin 48IU | Oxytocin 24IU/Placebo 24IU, Placebo 48IU, Oxytocin 48IU | Oxytocin 48IU, Oxytocin 24IU/Placebo 24IU, Placebo 48IU | Oxytocin 24IU/Placebo 24IU, Oxytocin 48IU, Placebo 48IU | Oxytocin 48IU, Placebo 48IU, Oxytocin 24IU/Placebo 24IU | Placebo 48IU, Oxytocin 48IU, Oxytocin 24IU/Placebo 24IU
Started | 1 | 2 | 2 | 1 | 1 | 1
Completed | 1 | 2 | 2 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third/Time 3 (1 Day at Week 3)
Arm/Group | Placebo 48IU, Oxytocin 24IU/Placebo 24IU, Oxytocin 48IU | Oxytocin 24IU/Placebo 24IU, Placebo 48IU, Oxytocin 48IU | Oxytocin 48IU, Oxytocin 24IU/Placebo 24IU, Placebo 48IU | Oxytocin 24IU/Placebo 24IU, Oxytocin 48IU, Placebo 48IU | Oxytocin 48IU, Placebo 48IU, Oxytocin 24IU/Placebo 24IU | Placebo 48IU, Oxytocin 48IU, Oxytocin 24IU/Placebo 24IU
Started | 1 | 2 | 2 | 1 | 1 | 1
Completed | 1 | 2 | 2 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Ten enrolled. One not randomized because on antipsychotic mediation at baseline. Nine started and one lost to follow-up after baseline. Eight participants were included in data analysis. Each participant received a dose of either 24IU oxytocin, 48IU oxytocin or placebo at each of 3 visits, spaced 1 wk apart, to the lab (i.e., baseline, wk 2, wk 3).
Groups:
- All Study Participants: Includes groups randomized to one of six different sequences of three interventions (placebo, oxytocin 24IU, oxytocin 48IU).
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.89 (4.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Eye Contact/Gaze During 10 Minute Social Challenge Task
Description: Number of times that eye gaze occurred (i.e., participant looked at female experimenter in the eyes) during 10 minute social challenge task (first 5 minutes social proximity, second 5 minutes social interaction). The social challenge task occurred 50 minutes after internasal dose (of placebo, placebo + oxytocin, or oxytocin) at baseline, week 2, and week 3 visits.
Time Frame: baseline, week 2, and week 3
Measure: Mean (Standard Error); unit: eye contact/gaze events per 10 minutes
Groups:
- Placebo: placebo (48IU)
- Oxytocin 24IU/Placebo 24IU: 24 international units of intranasal oxytocin and 24 international units of placebo
- 48IU OT: 48 international units of intranasal oxytocin
Arm/Group | Placebo | Oxytocin 24IU/Placebo 24IU | 48IU OT
Number analyzed (Participants) | 8 | 8 | 8
eye contact/gaze events per 10 minutes | 15.4 (3.5) | 20.9 (3.6) | 17.0 (4.5)

2. Secondary Outcome: Salivary Cortisol
Description: salivary cortisol level measured immediately before social challenge task and 20 minutes following social challenge task at each time point (i.e., baseline, week 2, and week 3)
Time Frame: baseline, week 2, and week 3
Measure: Mean (Standard Error); unit: nmol/L
Groups:
- Placebo: placebo (48 IU)
- 24IU OT: 24 international units of intranasal oxytocin and 24 IU of placebo
Arm/Group | Placebo | 24IU OT | 48IU OT
Number analyzed (Participants) | 8 | 8 | 8
nmol/L | 6.33 (.86) | 4.67 (.56) | 4.37 (.92)

ADVERSE EVENTS:
Groups:
- Intervention: Placebo 48IU: Two participants received placebo 48IU at baseline. Three participants received placebo 48IU at Time 2. Three participants received placebo 48IU at Time 3. This study is a cross-over design.
- Intervention: Oxytocin 24IU/Placebo 24IU: Three participants received Oxytocin 24IU/Placebo 24IU at baseline. Three participants received Oxytocin 24IU/Placebo 24IU at Time 2. Two participants received Oxytocin 24IU/Placebo 24IU at Time 3. This study is a cross-over design.
- Intervention: Oxytocin 48IU: Three participants received Oxytocin 48IU at baseline. Two participants received Oxytocin 48IU at Time 2. Three participants received Oxytocin 48IU at Time 3. This study is a cross-over design.
Arm/Group | Intervention: Placebo 48IU | Intervention: Oxytocin 24IU/Placebo 24IU | Intervention: Oxytocin 48IU
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 1/8 | 0/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention: Placebo 48IU (N=8) | Intervention: Oxytocin 24IU/Placebo 24IU (N=8) | Intervention: Oxytocin 48IU (N=8)
Bell's palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes